CLINICAL TRIAL: NCT02166359
Title: Effect of Extraneal (Icodextrin) on Triglyceride Levels in PD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, WON SUK AN, Professor, Dong-A University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXIT study
Record Dates: First submitted 2014-06-14; First posted 2014-06-18 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: End Stage Renal Disease
Keywords: Icodextrin; Triglyceride
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose group (Active Comparator): Glucose use of 2.5% or 4.25% dextrose solution at least 4 hours
  Interventions: Drug: Glucose solution
- Extraneal (Icodextrin) group (Experimental): Extraneal (Icodextrin) use at least 8 hours
  Interventions: Drug: Extraneal (Icodextrin)

INTERVENTIONS:
Drug: Extraneal (Icodextrin)
  Other Names: Extraneal; Icodextrin
  Arms: Extraneal (Icodextrin) group
Drug: Glucose solution
  Other Names: 2.5% dextrose solution; 4.25% dextrose solution
  Arms: Glucose group

SUMMARY:
Patients with chronic kidney disease (CKD) have a markedly higher prevalence of cardiovascular disease (CVD) than the general population. Dyslipidemia is considered a major cause of CVD in patients with CKD. Especially for peritoneal dialysis (PD) patients, the use of glucose as the osmotic agent in PD solutions has been associated with a variety of metabolic consequences ranging from acute hyperglycemia and hyperinsulinemia to dyslipidemia and weight gain. Among lipid abnormalities, hypertriglyceridemia is the most common in PD patients. A study showed that patients with high triglyceride levels were more insulin-resistant than those with normal triglyceride levels.

Insulin resistant is associated with atherogenic response represented high plasma levels of monocyte chemotactic protein-1 in a large cohort of dialysis patients. Therefore, high triglyceride level may play an important role to CV outcome of PD patients. PD solution decreasing triglyceride levels is essential in PD patients.

Icodextrin, a starch-derived high molecular weight glucose polymer was found to increase ultrafiltration compared to glucose solutions. Furthermore, a low peritoneal absorption of icodextrin, which is catabolized into maltose, considerably reduces caloric uptake. Therefore, icodextrin may have an additional favorable effect on triglyceride level.

There are several studies regarding the effect of icodextrin on triglyceride level in PD patients. However, the outcomes are controversial, some studies showed no association between icodextrin and triglyceride change, even the others showed positive results but these also have study design limitations such as non-randomized study or secondary primary outcome. It is not clear about the effect of icodextrin on triglyceride especially in PD patients without diabetes.

The investigators therefore want to conduct a randomized, cross-over, controlled multicenter trial comparing icodextrin solution and glucose solution in PD patients with and without diabetes, focusing on triglyceride change.

ELIGIBILITY:
Inclusion Criteria:

* PD patients agree with written informed consent
* Incident and prevalent PD patients on dialysis for at least 3month
* PD patients treated with two glucose solutions including 2.5% or 4.25% dextrose solution at least 4hour

Exclusion Criteria:

* PD patients with allergy to starch-based polymers
* PD patients with glycogen storage disease
* PD patients with maltose or isomaltose intolerance
* PD patients with active alcohol/substance abuse
* Pregnant or nursing PD patients
* PD patients with an episode of peritonitis and active systemic infection within 4weeks before study initiation
* PD patients newly prescribed with lipid-lowering medications, including statins, omega-3 fatty acids or sevelamer hydrochloride within 3 months before randomization
* PD patients with triglyceride level> 500 mg/dL/L or <100 mg/dL
* PD patients with albumin level < 3.0 gram/dL
* PD patients treated with automated PD
* PD patients had been treated or are treating with icodextrin PD solutions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The mean difference and change of triglyceride levels after follow up between 2 groups | baseline and 3 months after intervention
  The difference and change of triglyceride after follow up between 2 groups (glucose group with diabetes (n=20) vs. icodextrin group with diabetes (n=20) and glucose group without diabetes (n=20) vs. icodextrin group without diabetes (n=20) )

SECONDARY OUTCOMES:
The mean difference and change of erythrocyte membrane monounsaturated fatty acid content and oleic acid content | baseline and 3 months after intervention
The mean difference and change of total cholesterol , LDL, HDL, very low-density lipoprotein, apolipoprotein A and apolipoprotein B | baseline and 3 months after intervention
The mean difference and change of blood glucose level, insulin and HbA1c | baseline and 3 months after intervention
The mean difference and change of ultrafiltration volume | baseline and 3 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University Hospital, Busan, South Korea